CLINICAL TRIAL: NCT06665945
Title: The SENTRY Study: Testing Whether Changes in Platelet RNA Enhance the Early Diagnosis of Ovarian Cancer
Acronym: SENTRY
Status: Recruiting | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: HCI175150
Record Dates: First submitted 2024-09-11; First posted 2024-10-30 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — This study will obtain platelet RNA samples from whole blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Women with a Recent Diagnosis of Ovarian Cancer (n=90)
  Interventions: Diagnostic Test: Platelet RNA expression
- Women with a Recent Diagnosis of Ovarian Mass (n=125)
  Interventions: Diagnostic Test: Platelet RNA expression
- Control Women without Ovarian Cancer (n=30)
  Interventions: Diagnostic Test: Platelet RNA expression

INTERVENTIONS:
Diagnostic Test: Platelet RNA expression — The SENTRY (Stability Enhanced Transcriptional Analytics) Study is to test whether combining a unique analytical approach with changes in platelet RNA expression accurately diagnoses ovarian cancer.

SUMMARY:
The purpose of the SENTRY (Stability Enhanced Transcriptional Analytics) Study is to test whether combining a unique analytical approach with changes in platelet RNA expression accurately diagnoses ovarian cancer. Using retrospective data, the investigators have developed an approach that appears to accurately classify ovarian cancer with relatively high sensitivity and specificity. The SENTRY Study will build upon these retrospective analyses to prospectively recruit women with ovarian cancer or an ovarian mass (and healthy control women), obtain platelet RNA samples from whole blood, and perform validation analyses to test our hypothesis.

ELIGIBILITY:
Study Population 1: Women with a Recent Diagnosis of Ovarian Cancer (n=90)

Inclusion Criteria:

1. Women aged 21 years or older
2. Diagnosed with any stage or type of ovarian cancer within the last 8 weeks

Exclusion Criteria:

1. Any other active malignancy
2. Other diagnosis of any cancer within the last 6 months
3. Treatment for any cancer within the last 6 months
4. History of ovarian cancer at any time
5. Currently receiving chemotherapy for ovarian cancer
6. Has already undergone complete ovarian mass resection
7. Unable to provide blood sample

Study Population 2: Control Women without Ovarian Cancer (n=30)

Inclusion Criteria:

1. Women aged 21 years or older

Exclusion Criteria:

1. Any active malignancy or diagnosis of cancer within the last 6 months
2. Treatment for any cancer within the last 6 months
3. Hospitalization or surgery (other than minor surgery such as mole removal) within the last 8 weeks
4. Renal failure (defined as eGFR < 60 mL/min/1.73m² or on dialysis)
5. Liver failure (defined as having hepatic encephalopathy of any degree, OR moderately severe coagulopathy defined as INR ≥ 1.5, OR known cirrhosis, OR ALT of ≥ 10X ULN, OR total bilirubin of ≥ 3.0 mg/dL, OR diagnosis of liver failure)
6. Decompensated or end-stage heart failure (defined as ACC/AHA Stage C or Stage D heart failure)
7. Poorly controlled diabetes mellitus (defined as a HbA1c > 9.0%)
8. Venous thrombosis, myocardial infarction, or stroke within the last 8 weeks
9. Currently pregnant or have been pregnant within the last 12 weeks
10. Any blood product transfusion within the last 8 weeks
11. Personal history of ovarian cancer at any time
12. History of bilateral salpingo-oophorectomy
13. History of oophorectomy
14. Unable to provide blood sample

Study Population 3: Women with a Recent Diagnosis of Ovarian Mass (n=125)

Inclusion Criteria:

1. Women aged 21 years or older
2. Diagnosed with any type of ovarian mass within the last 8 weeks

Exclusion Criteria:

1. Any diagnosis of active malignancy
2. Any diagnosis of any cancer within the last 6 months
3. Treatment for any cancer within the last 6 months
4. History of ovarian cancer at any time
5. Currently receiving chemotherapy for ovarian cancer
6. Has already undergone complete ovarian mass resection
7. Unable to provide blood sample

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be patients in the Huntsman Cancer Hospital Clinics in Salt Lake City, Utah.
Sampling Method: Non-Probability Sample
Enrollment: 245 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Early-Stage Ovarian Cancer Detection | Following informed consent (study visit 1, day 1).
  The goal is to determine if changes in platelet RNA expression accurately diagnoses ovarian cancer. This outcome will report the number of true positive, true negative, false positive, and false negative results from this assay.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Werner, MD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No